CLINICAL TRIAL: NCT06130462
Title: Detection of Aluminium-reactive T-lymphocytes in Patients With Vaccination Granulomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Allergy Research Center, Denmark (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: H-20073116
Record Dates: First submitted 2023-11-08; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Granuloma; Aluminum Allergy
Keywords: aluminum; allergy; contact dermatitis; vaccination granuloma; LPT; SCIT
MeSH Terms: conditions — Granuloma; Hypersensitivity; Dermatitis, Contact

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LPT aluminium (Active Comparator): Investigation of participants with aluminium allergy versus healthy controls. Aluminium in different concentrations are added to the blood samples to elicit a response
  Interventions: Diagnostic Test: Aluminum
- LPT control (Placebo Comparator): Tetanus toxoid was added to blood samples as control substance.
  Interventions: Diagnostic Test: Tetanus toxoid

INTERVENTIONS:
Diagnostic Test: Aluminum — Different concentrations of aluminium added to the blood test in vitro
  Arms: LPT aluminium
Diagnostic Test: Tetanus toxoid — Used as control substance
  Arms: LPT control

SUMMARY:
Vaccines and subcutanoeus immunotherapy vaccines often contains aluminium, and may induce itching granulomas at the injection site. This is usually diagnosed by patch testing. Another way of detecting metal allergy is by investigation metal-specific cells in the blood.

We include participants both with and without granulomas, all have a blood test taken where we investigate if any participants have aluminium-specific cirkulation cells, and whether we can detect a difference between participants with and without granulomas.

DETAILED DESCRIPTION:
Aluminium-adsorbed vaccines and subcutaneous immunotherapy may induce vaccination granulomas at injection site. Most children have concormitant aluminium contact allergy diagnosed by path testing, but in adults the allergy can rarely be detected by patch tests.

An alternative to patch testing is the blood in vitro lymphocyte proliferation test (LPT), which we investigated using a well-established LPT protocol. This has previously been shown to detect and characterize metal-specific cells and was used to detect circulating aluminium-specific proliferation. The LPT test is based on a single blood sample and has mostly been used to detect drug hypersensitivity. Still, its role in detecting metal allergy is expanding, with recent studies suggesting using the test as a supplement to the patch test when only a few allergens are to be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Indivicuals with vaccination granulomas
* controls without granulomas and no suspected contact allergies

Exclusion Criteria:

* pregnancy, breastfeeding, recent vaccination, skin diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
LPT | 7 days
  Proliferation of T-cells

CONTACTS AND LOCATIONS:
Overall Officials: Lars Blom, PhD, Study Director — Allergy clinic, Gentofte Hospital
Locations (1):
- National Allergy Research Centre, Gentofte Hospital, Hellerup, Denmark